CLINICAL TRIAL: NCT03256162
Title: Ketamine as an Adjunctive Therapy for Major Depression - a Randomised Controlled Pilot Trial: The KARMA-Dep Trial
Brief Title: Ketamine as an Adjunctive Therapy for Major Depression
Acronym: KARMA-dep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St Patrick's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Prof Declan McLoughlin, Professor, St Patrick's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 01/17; 2016-004764-18 (EudraCT Number)
Record Dates: First submitted 2017-08-02; First posted 2017-08-21 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Episode; Unipolar Depression; Bipolar Depression
Keywords: ketamine; glutamate
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants will receive four once-weekly infusions of ketamine at 0.05mg/kg. All infusions will be administered by a consultant anaesthetist.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Participants will receive four once-weekly infusions of midazolam at 0.045mg/kg. All infusions will be administered by a consultant anaesthetist.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — A sub-anaesthetic dose of ketamine will be administered in four infusions, each one week apart.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Midazolam — A sub-anaesthetic dose of midazolam will be administered in four infusions, each one week apart.
  Other Names: Hypnovel
  Arms: Midazolam

SUMMARY:
Randomised, controlled, parallel-group, pilot clinical trial of ketamine vs. midazolam as an adjunctive therapy for depression. The main purpose of the pilot study is to assess trial processes to help inform a future definitive trial.

DETAILED DESCRIPTION:
Pragmatic, randomised, controlled, parallel-group, pilot trial. Trial participants will be patients admitted to St Patrick's University Hospital for treatment of a depressive episode. The investigators aim to recruit up to 20 participants who will be eligible for this study and randomly allocate 10 patients to each group. The participants will undergo usual inpatient care as prescribed by their treating team for the index acute depressive episode. Both participants and assessors will be blind to treatment allocation. Consented participants will be randomly allocated in a 1:1 ratio to a four week course of either once-weekly ketamine or midazolam infusions. Block randomisation will be independently performed. Physical, psychotomimetic and cognitive outcomes will be monitored before, during and after infusions. Blood samples will be taken at four time-points in the first infusion session and before the final infusion for neuroplasticity biomarker studies. Both groups will continue treatment as usual. Participates will also be followed up over a three month period.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Hamilton Rating Scale for Depression-24 item version (HRSD-24) score of ≥21
* Voluntary admission for treatment of an acute depressive episode
* Meet Diagnostic and Statistical Manual of Mental Disorders , Fifth Edition (DSM-V) criteria for a major depressive disorder (MDD) and bipolar affective disorder (current episode depression)

Exclusion Criteria:

* Current involuntary admission
* Medical condition rendering unfit for ketamine/midazolam
* Active suicidal intention
* Dementia
* History of Axis 1 diagnosis other than major depression
* Electroconvulsive Therapy (ECT) administered within the last two months
* Alcohol/substance dependence in previous six-months
* Pregnancy or inability to confirm use of adequate contraception during the trial
* Breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Declan M McLoughlin, PhD, Principal Investigator — St Patrick's Mental Health Services and Trinity College Dublin
Locations (1):
- St Patrick's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallagher B, Foley M, Slattery CM, Gusciute G, Shanahan E, McLoughlin DM. Ketamine as an adjunctive therapy for major depression - a randomised controlled pragmatic pilot trial (Karma-Dep Trial). HRB Open Res. 2022 Jan 27;3:90. doi: 10.12688/hrbopenres.13182.2. eCollection 2020. PMID 35036831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were those who were admitted to St Patrick's University Hospital, Dublin, for treatment of a major depressive episode (either unipolar or bipolar depression) between 06.09.17 and 12.06.18.
Pre-assignment Details: Treatment-as-usual, by the participants' treating teams, continued throughout the entire trial.
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 13 | 12
Completed | 8 | 8
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (13.1) | 52.3 (12.5) | 50.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
The Hamilton Rating Scale for Depression-24 Item Version (HRSD-24) [Mean (Standard Deviation); unit: units on a scale] — The HRSD assesses severity of depressive symptoms and is commonly used to measure depression severity. It was initially a 17-item format with the optional addition of 4 items making up the 21-item version. In addition to the original 21 items, the 24-item HRSD includes items on helplessness, hopelessness and worthlessness; its score range is 0-77, with higher scores reflecting greater burden of depressive symptoms.
  units on a scale | 28.4 (4.3) | 27.4 (4.3) | 27.7 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: The Hamilton Rating Scale for Depression-24 Item Version (HRSD-24)
Description: The HRSD assesses severity of depressive symptoms and is commonly used to measure depression severity. It was initially a 17-item format with the optional addition of 4 items making up the 21-item version. In addition to the original 21 items, the 24-item HRSD includes items on helplessness, hopelessness and worthlessness; its score range is 0-77, with higher scores reflecting greater burden of depressive symptoms.
  Response to antidepressant treatment is defined as achieving ≥60% decrease from baseline HRSD-24 and score ≤16. Remission criteria are ≥60% decrease in HRSD from baseline and score ≤10. Criteria for relapse are ≥10 point increase in HRSD-24 compared to responder baseline score plus HRSD ≥16; in addition, increase in the HRSD should be maintained one week later.
  Participants will have a baseline (T0) HRSD-24 score. This will be repeated 1 week after each of 4 once-weekly infusions (T1-4) and follow-up measures after another 5 (T9) and 11 (T15) weeks, week 15 is reported.
Time Frame: 15 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
score on a scale | 11.2 [6.2 to 16.2] | 16.6 [7.8 to 25.3]

2. Secondary Outcome: The Quick Inventory of Depressive Symptoms, Self-report Version (QIDS-SR16)
Description: The QIDS-SR16 is a validated self-report measure of depressive symptoms. This consists of 16 questions rated 0-3. Its score range is 0-48, with higher scores reflecting greater burden of depressive symptoms.
  Participants will have a baseline (T0) QIDS-SR16 score. This will be repeated one week after each of four once-weekly infusions (T1-4) and follow-up measures after another five (T9) and 11 (T15) weeks. Week 15 scores are reported.
Time Frame: 15 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
score on a scale | 9.1 [5.6 to 12.6] | 11.4 [4.9 to 18.0]

3. Secondary Outcome: The Clinician-Administered Dissociative States Scale (CADSS)
Description: The CADSS measures dissociative symptoms. It will be administered before, during and after infusions in order to capture the range of possible subjective side effects of either agent. This consists of 23 questions and scores for each question range from 0-4. The maximum score is 92 with higher scores indicating more dissociative symptoms.
  Participants will have the CADSS performed before, during (+30mins) and after (+60mins) each of the four once-weekly infusions.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
score on a scale | 5.3 (7.2) | 2.5 (3.5)

4. Secondary Outcome: The Brief Psychiatric Rating Scale (BPRS)
Description: The BPRS measures psychotomimetic effects. The investigators will use the positive symptoms subscale of the Brief Psychiatric Rating Scale. The 4-item positive symptoms subscale measures suspiciousness, hallucinations, unusual thought content, and conceptual disorganisation. Each question is scored between 0-7. The maximum score in this 4-item questionnaire is 28. Higher scores indicate more severe psychotic symptoms.
  Participants will have the BPRS performed before, during (+30mins) and after (+60mins) each of the four once-weekly infusions.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
score on a scale | 4.1 (0.4) | 4.0 (0)

5. Secondary Outcome: Young Mania Rating Scale (YMRS; Mood Item)
Description: Investigators will use the mood item of them YMRS to assess for psychotomimetic effects. This item is rated 0-4. The higher scores reflect elevated mood.
  Participants will have the YMRS performed before, during (+30mins) and after (+60mins) each of the four once-weekly infusions.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
score on a scale | 0.1 (0.4) | 0.1 (0.4)

6. Secondary Outcome: The Patient-Rated Inventory of Side Effects (PRISE)
Description: The PRISE will be used to document other general adverse events by patients before, during and after infusions. This is a patient self-report used to qualify side effects by identifying and evaluating the tolerability of each symptom. It is a 9 item assessment of the side effects in the following symptom domains; Gastrointestinal, Heart, Skin, Nervous System, Eyes/Ears, Genital/Urinary, Sleep, Sexual Functioning, and Other. Each domain has multiple symptoms which can be endorsed. For each domain the patient rates whether or not the symptoms are tolerable or distressing. Data below represent the number of participants from which there was an endorsement of each listed event.
  Participants will have the PRISE performed before, during (+30mins) and after (+60mins) each of the four once-weekly infusions.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
participants
  dry mouth | 1 | 1
  diarrhoea | 0 | 0
  Constipation | 0 | 0
  Nausea / vomiting | 0 | 0
  Palpitation | 0 | 0
  Chest pain | 0 | 0
  Rash | 0 | 0
  Headache | 0 | 0
  Tremors | 0 | 0
  Poor coordination | 1 | 0
  Dizziness | 2 | 0
  Blurred vision | 0 | 0
  Difficulty urinating | 0 | 0
  Difficulty sleeping | 0 | 0
  Sleeping too much | 0 | 1
  Anxiety | 2 | 0
  Poor concentration | 0 | 1
  Restlessness | 2 | 0
  Fatigue | 3 | 1

7. Secondary Outcome: The Montreal Cognitive Assessment (MoCA)
Description: The MOCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, conceptual thinking, calculations, and orientation. It is scored out of a maximum of 30. The higher scores indicate better cognition.
  The MOCA will be performed at baseline, one day after infusions 1 and 4 and 12 weeks after the final infusion.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 8 | 8
score on a scale | 26.4 (3.1) | 28.5 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected over the entire study time frame, 10 months (September 2017 - June 2018). For each participant, data was collected over a period of 15 weeks which included 3 weeks of intervention and 12 weeks of follow up assessments.
Description: Tolerability of the trial agents was assessed at multiple points before, during and after treatment sessions using various assessments including the CADSS, BPRS, PRISE and YMRS. These have been used in other clinical trials which have used ketamine as a treatment for depressive disorders. We also carried out physical health assessments during the infusion clinics (e.g. vital signs).
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

LIMITATIONS AND CAVEATS:
As this is a pilot trial, participant numbers are low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03256162/Prot_SAP_000.pdf